CLINICAL TRIAL: NCT03368937
Title: The International Diabetes Closed Loop (iDCL) Trial: Clinical Acceptance of the Artificial Pancreas - A Pilot Test of t:Slim X2 With Control-IQ Technology
Brief Title: A Pilot Test of t:Slim X2 With Control-IQ Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20251; UC4DK108483 (NIH)
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Results first posted 2019-02-27 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Artificial Pancreas (AP); Closed Loop Control (CLC); Continuous Glucose Monitor (CGM); Insulin Pump

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Tandem t:slim X2 with Control-IQ Technology (Experimental): Subjects will use the Tandem t:slim X2 with Control-IQ Technology during a 36-48 hour hotel admission.
  Interventions: Device: Tandem t:slim X2 with Control-IQ Technology

INTERVENTIONS:
Device: Tandem t:slim X2 with Control-IQ Technology — Subjects will wear the Tandem t:slim X2 with Control-IQ Technology during a 36-48 hour hotel admission.

SUMMARY:
A 36-48 hour admission testing the t:slim X2 with Control-IQ Technology

DETAILED DESCRIPTION:
The objective of the study is for clinical staff to gain experience using the proposed artificial pancreas system named t:slim X2 with Control-IQ Technology and assess usability in a supervised setting prior to initiating home use in a Training protocol.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, a subject must meet the following criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year
2. Use of an insulin pump for at least 6 months with established parameters for basal rate(s), carbohydrate ratio(s) and insulin sensitivity factor(s) for at least 3 months.
3. Age 18.0 to <75.0 years
4. Hemoglobin A1c <10.5%
5. For females, not currently known to be pregnant If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a subject in the study. A negative serum or urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study. Also, subjects who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
6. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
7. Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol
8. Currently using no insulins other than one of the following rapid-acting insulins at the time of enrollment: insulin lispro (Humalog), insulin aspart (Novolog), or insulin glulisine (Apidra). Willingness to switch to lispro (Humalog) or aspart (Novolog) if using glulisine (Apidra).
9. Total daily insulin dose (TDD) at least 10 U/day and ≤100 U/day
10. Weight at least 25 kg and not greater than 140 kg

Exclusion Criteria:

1. More than one episode of diabetic ketoacidosis (DKA) in the 6 months prior to enrollment
2. More than one episode of severe hypoglycemia involving seizure or loss of consciousness in the 6 months prior to enrollment
3. Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals).
4. Hemophilia or any other bleeding disorder
5. A condition, which in the opinion of the investigator or designee, would put the subject or study at risk
6. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
7. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc. or TypeZero Technologies, LLC, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue A Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brown S, Raghinaru D, Emory E, Kovatchev B. First Look at Control-IQ: A New-Generation Automated Insulin Delivery System. Diabetes Care. 2018 Dec;41(12):2634-2636. doi: 10.2337/dc18-1249. Epub 2018 Oct 10. PMID 30305346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tandem t:Slim X2 With Control-IQ Technology
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tandem t:Slim X2 With Control-IQ Technology
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: System Suitability
Description: Technology Acceptance Questionnaire Score Scores are on a Likert Scale of 1-Not at All to 5-Extremely for Ease of Use, Usability and Trust in System Scores.
Time Frame: 36-48 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Tandem t:Slim X2 With Control-IQ Technology
Number analyzed (Participants) | 5
score on a scale
  Ease of Use | 5 [5 to 5]
  Usefulness | 4.8 [4 to 5]
  Trust in System | 5 [5 to 5]

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Tandem t:Slim X2 With Control-IQ Technology
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03368937/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03368937/ICF_001.pdf